CLINICAL TRIAL: NCT02145312
Title: An Open Label, Single Arm, Multicenter Phase II Study of BYL719 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck Who Failed to Respond to Platinum-based Therapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0147
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Recurrence | interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BYL719 (Experimental): BYL719 is an oral class I α-specific PI3K inhibitor belonging to the 2-aminothiazole class of compounds.
  Interventions: Drug: BYL719

INTERVENTIONS:
Drug: BYL719 — BYL719 is an oral class I α-specific PI3K inhibitor belonging to the 2-aminothiazole class of compounds.

SUMMARY:
One promising approach to the treatment of cancer is inhibition or modulating the crucial signal transduction pathway of PI3K-Akt-mTOR. Several PI3K inhibitors are being tested in the clinical trials for cancer treatment but not for the head and neck cancer yet. BYL719 is an alpha specific I PI3K inhibitor. It showed significant, concentration dependent cell growth inhibition and induction of apoptosis. We suggest multicenter single arm phase II study to determine anti-tumor effects of BYL719 in patients with recurrent and/or metastatic SCCHN who failed to prior chemotherapy regimens. Enrollment will be done in 5 or more clinical trial centers in Korea. Primary objective is to evaluate disease control rate (DCR) at 8 weeks of BYL719, and the efficacy will be evaluated by the investigators analysis based on RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent or metastatic squamous-cell carcinoma of head and neck (SCCHN), except nasopharyngeal carcinoma
2. 18 years of age or older
3. Patients must have progressive disease after one or two prior chemotherapy regimens including platinum-based chemotherapy given for the treatment of recurrent and/or metastatic disease, or within 6 months after concurrent chemoradiation (with or without induction chemotherapy) given as a definitive treatment.
4. Life expectancy of at least 12 weeks
5. Ineligibility for local therapy (surgery or radiation for curative intent)
6. At least one lesion that is measurable according to the RECIST 1.1 criteria by CT or MRI
7. ECOG performance score of 0-2
8. Availability of tissue samples (archival tissue or rebiopsied tissues) for molecular analysis (representative paraffin block or unstained sections from tumor diagnostic specimen are mandatory)
9. Adequate organ function and laboratory parameters as defined by:

   * Absolute neutrophil count (ANC) ≥1.5x109/L
   * Hemoglobin (Hgb) ≥ 9 g/dl (which may be reached by transfusion)
   * Platelets (PLT) ≥ 100 x 109/L (which may be reached by transfusion)
   * AST/SCOT and ALT/SGPT ≤ 2.5xULN (upper limit of normal) or ≤ 5 x ULN if liver metastases are present
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum creatinib ≤ 1.5 x ULN or calculated or directly measured CrCl ≥ 50% LLN (lower limit of normal)
   * Fasting plasma glucose (FPG) < 140 mg/dL/7.8mmol/L

Exclusion Criteria:

1. Prior treatment with PI3K pathway inhibitors
2. Nasopharyngeal carcinoma
3. Uncontrolled, untreated brain metastasis. Patients with treated/controlled and asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases ≥ 28 days (must include radiotherapy and/or surgery) and, if on corticosteroid therapy, should be receiving a stable low dose (e.g. dexamethasone 4 mg or equivalent dose of another corticosteroid for at least 14 days before start of study treatment).
4. Surgery, chemotherapy or irradiation within 3 weeks of study entry
5. Concomitant chemotherapy, hormonal therapy or immunotherapy
6. Clinically significant cardiac disease or impaired cardiac function, such as:

   * Congestive heart failure (CHF) requiring treatment (New Yort Heart Association (NYHA) Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO), or uncontrolled arterial hypertension defined by blood pressure > 140/100 mmHg at rest (average of 3 consecutive readings)
   * History or current evidence of clinically significant cardiac arrhythmias, arterial fibrillation and/or conduction abnormality, e.g. congenical long QT syndrome, high grade/complete AV-blockage
   * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening
   * QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening ECG
7. Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with FPG ≥ 140 mg/dL/7.8mmol/L, or history of documented steroid-induced diabetes mellitus.
8. Patient who cannot take the oral drug
9. Impaired GI function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
10. Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment.
11. Previous or concomitant malignant disease, except adequately treated basal cell cancer of the skin or cervical cancer in situ, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior study entry
12. Pregnant woman, Breast-feeding woman
13. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial (infection/inflammation, intestinal obstruction, social/psychological complications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 8 weeks of BYL 719 administered as therapy
  The primary objective of this study is to evaluate disease control rate (DCR) at 8 weeks of BYL719 administered as therapy for patient with recurrent/metastatic head and neck squamous cell carcinoma, comparing with historical control. Efficacy evaluation will be based on RECIST version 1.1. DCR will be expressed percent and 95% confidence interval.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 24 months
Progression-free survival (PFS) | 24 months
Overall survival (OS) | 24 months
Time to progression (TPP) | 24 months
Drug toxicity and safety analysis | 24 months
Quality of life assessment | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea